CLINICAL TRIAL: NCT04403321
Title: Efficacy and Safety of Eltrombopag + Tacrolimus in Chinese Refractory or Relapsed Aplastic Anemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELT-1
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Aplastic Anemia; Drug Effect
MeSH Terms: conditions — Anemia, Aplastic | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Placebo Comparator): Eltrombopag and the placebo would be applied. Eltrombopag will be started at 25 mg/day and increased by 25 mg/day every 2 weeks according to the platelet count up to 150 mg/day, or the best response was achieved.
  Interventions: Drug: Placebo (for Tacrolimus)
- Eltrombopag + Tacrolimus (Experimental): Eltrombopag and tacrolimus would be applied. Eltrombopag will be started at 25 mg/day and increased by 25 mg/day every 2 weeks according to the platelet count up to 150 mg/day, or the best response was achieved. Tacrolimus will be given at 1mg bid with the target trough concentration of 4-10 ng/mL throughout the study.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus will be given at 1mg bid with the target trough concentration to be 4-10 ng/mL.
  Other Names: experimental
  Arms: Eltrombopag + Tacrolimus
Drug: Placebo (for Tacrolimus) — placebo will be given at 1mg bid.
  Other Names: control
  Arms: Eltrombopag

SUMMARY:
This is a randomized, open-label, phase II study to compare the efficacy of eltrombopag combined with tacrolimus to eltrombopag alone in Chinese subjects with refractory or relapsed aplastic anemia. The safety would also be evaluated. Patients would be randomized to receive eltrombopag alone or eltrombopag combined with tacrolimus. Treatment with eltrombopag will be started at 25 mg/day and increased by 25 mg/day every 2 weeks according to the platelet count up to 150 mg/day, or the best response was achieved. Tacrolimus will be given at 1mg bid with the target trough concentration of 4-10 ng/mL throughout the study. The hematological response rate and safety will be recorded and compared at 3, 6 months and 1 year after starting the study treatment (Week 13, 26 and 52).

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a previous diagnosis of aplastic anemia and had no response or relapsed following at least one treatment course in a period time of ≥ 6 months of immunosuppression containing CsA or CsA+anti-thymocyte globulin (ATG);
2. Current diagnosis of aplastic anemia by bone marrow biopsy;
3. did not receive HSCT nor were HSCT candidates;
4. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
5. Patient with QTcF (Fridericia's QT correction formula) at screening <450 msec, or <480 msec with bundle branch block, as determined via the mean of a triplicate ECG and assessed at site.
6. Subjects are able to understand and comply with protocol requirements and instructions and have signed and dated informed consent.

Exclusion Criteria:

1. Congenital aplastic anemia;
2. Presence of chromosomal aberration;
3. Evidence of a clonal hematologic bone marrow disorder on cytogenetics;
4. Have any concomitant malignancies and must be fully recovered from treatment for any other malignancy and have been disease-free for 5 years;
5. AST or ALT ≥3 times the upper limit of normal;
6. Serum creatinine, total bilirubin, or alkaline phosphatase >1.5 x ULN;
7. Cardiac disorder (NYHA) functional classification Grade II/III/IV;
8. Past history of thromboembolic event (including anti-phospholipid antibody syndrome) and current use of anticoagulants;
9. Infection not adequately responding to appropriate therapy;
10. Other known or suspected underlying primary immunodeficiency;
11. Prior treatment with eltrombopag, romiplostim, or any other TPO (thrombopoietin) receptor agonist;
12. Pregnant or nursing (lactating) woman;

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
ORR at 6 Months | Week 26
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR) at Week 26

SECONDARY OUTCOMES:
ORR at 3 Months | Week 14
  ORR will be calculated after 3 months of treatment by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Changes in Haemoglobin in the Absence of Red Blood Cells Transfusion | Week 26
  The change in hematology values ( haemoglobin) were evaluated
Changes in Platelet in the Absence of Platelet Transfusion | Week 26
  The change in hematology values (platelet) were evaluated
Duration of hematologic response | by 6 months (all patients), at 24 months (responders only)
  Time from the date of the start of the first response to the date of first relapse defined as again meeting criteria for aplastic anemia
Percentage of patients with clonal evolution to myelodysplasia, PNH, acute leukemia | 12 months
  Clonal evolution to myelodysplasia is defined as a new marrow cytogenic abnormality with or without characteristic dysplastic marrow findings. Evolution to leukemia is defined as greater than 20% peripheral blood and/or marrow blasts. Evolution to paroxysmal nocturnal hemoglobinuria (PNH) is defined as a clone at baseline < 10% that rose to greater than 50% on study.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: email request